CLINICAL TRIAL: NCT05355467
Title: Efficacy and Safety of Ricovir® in Maintaining Durability of Viral Response in Chronic Hepatitis B Patients Who Have Been Treated With Viread® and Have Undetectable HBV DNA in Serum
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Mylan (Taiwan) Ltd (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Mylan-Ricovir-TW-01
Record Dates: First submitted 2022-04-25; First posted 2022-05-02 (Actual); Last update posted 2022-05-02 (Actual); Status verified 2022-04

CONDITIONS: Chronic Hepatitis B Infection
MeSH Terms: conditions — Hepatitis B, Chronic | interventions — Tenofovir

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Ricovir® group (Experimental)
  Interventions: Drug: Tenofovir disoproxil fumarate
- Historical Control Group (Other)
  Interventions: Other: Historical Data

INTERVENTIONS:
Drug: Tenofovir disoproxil fumarate — Ricovir® (tenofovir disoproxil fumarate 300 mg) 1 tablet daily. The overall treatment period is 24 weeks.
  Arms: Ricovir® group
Other: Historical Data — Historical Data
  Arms: Historical Control Group

SUMMARY:
This is a phase IV, open label, historical controlled comparative study to evaluate the efficacy and safety of Ricovir® in maintaining durability of viral response in CHB patients who have been treated with Viread® and have undetectable HBV DNA in serum by real-time polymerase chain reaction (PCR) assay.

ELIGIBILITY:
Ricovir® Group

Inclusion Criteria:

* Male or female aged more than 20 years old;
* CHB patients who have been treated with Viread® for more than 1 year;
* Serum HBV DNA level is undetectable (not detected or <20 IU/mL) at screening;
* Informed consent must be obtained before the commencement of any screening procedures or study drugs

Exclusion Criteria:

* Patients with active HCC or other types of malignancy;
* Patients with impaired renal function (defined as eGFR ≦ 30 mL/min/1.73m2);
* Patients with hepatitis A (HAV), hepatitis C (HCV), hepatitis D (HDV) or human immunodeficiency virus (HIV) coinfection;
* Patients with alcohol dependence or addiction;
* Patients with autoimmune hepatitis;
* Patients with primary biliary cholangitis (PBC);
* Pregnancy, planning on getting pregnant, or breast-feeding;
* History of allergy, hypersensitivity, intolerance, or experiencing severe adverse reactions to tenofovir or any ingredient of the study drug;
* Not suitable for participating in this trial at the investigator's discretion.

Historical Control Group

Eligible individuals will be obtained from the TCVGH historical database based on matching (1:1) in terms of age (±5 years) and gender. To be eligible for the study, subjects must meet all of the following criteria:

* Male or female aged more than 20 years old;
* CHB patients who had been treated with Viread® for more than 1 year;
* Patients who had discontinued Viread® therapy for at least 24 weeks during the period from January 2014 to December 2021 and had undetectable HBV DNA (not detected or <20 IU/mL) in serum at the time of discontinuation;
* Patients who have the data of HBV DNA level 24 weeks after the time of discontinuation, with a time window of +4 weeks is allowed;
* The informed consent requirement will be waived based on the approval of IRB.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2019-08-21 (Actual); Primary Completion 2021-07-13 (Actual); Study Completion 2021-07-13 (Actual)

PRIMARY OUTCOMES:
Assessment of the rates of virological recurrence of HBV | Week 24
  To assess the rates of virological recurrence of HBV at Week 24 with Ricovir® treatment.

SECONDARY OUTCOMES:
Comparison of the HBV DNA levels between Ricovir® group and historical control group | Week 24
  To compare the HBV DNA levels at Week 24 between Ricovir® group and historical control group.
Comparison of the rates of virological recurrence of HBV between Ricovir® group and historical control group. | Week 24
  To compare the rates of virological recurrence of HBV at Week 24 between Ricovir® group and historical control group.
Monitoring of Safety profile for subjects in Ricovir® group | Up to 24 weeks
  For subjects in Ricovir® group, physical examination, vital signs, HBV DNA level, and concomitant medications will be evaluated at Week 4, 12 and 24 after treatment. Hematology and clinical biochemistry will be performed every 12 weeks. Adverse events (AEs) will be monitored continuously during the study.

CONTACTS AND LOCATIONS:
Overall Officials: Sanjay Hadigal, Dr., Study Director — Mylan Pharmaceuticals Private Limited
Locations (1):
- Taichung Veterans General Hospital, Taichung, Taiwan